CLINICAL TRIAL: NCT06342622
Title: Application of Artificial Intelligence for Young-onset Colorectal Cancer Screening Based on Electronic Medical Records
Brief Title: Young-onset Colorectal Cancer Screening Based on Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: Weiguo Dong
Record Dates: First submitted 2024-03-15; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: Young-onset colorectal cancer; Cancer screening; Artificial intelligence; Machine learning
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with young-onset colorectal cancer: Patients were diagnosed with young-onset colorectal cancer after receiving colonoscopy examination.
  Interventions: Diagnostic Test: Using routine clinical data and machine learning models.
- Patients without young-onset colorectal cancer: Patients were ruled out young-onset colorectal cancer after receiving colonoscopy examination.
  Interventions: Diagnostic Test: Using routine clinical data and machine learning models.

INTERVENTIONS:
Diagnostic Test: Using routine clinical data and machine learning models. — This study used clinical data and machine learning model to screen young-onset colorectal cancer.

SUMMARY:
In this study, we aimed to develop, internally and temporally validate the machine learning models to help screen YOCRC bansed on the retrospective extracted Electronic Medical Records (EMR) data.

DETAILED DESCRIPTION:
Diagnosis of young-onset colorectal cancer (YOCRC) has become more common in recent decades. Screening CRC among younger adults still remains a challenge. In this study, We plan to retrospectively extracte the relevant clinical data of young individuals who underwent colonoscopy from 2013 to 2022 using Electronic Medical Record (EMR). Multiple supervised machine learning techniques will be applied to distinguish YOCRC and non-YOCRC individuals, the above classifiers will be trained and internally validated in the training dataset and internal validation dataset admitted between 2013 and 2021, respectively. We will also assess the temporal external validity of the classifiers based on the admissions from 2022.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with CRC (YOCRC group)
* Age at 18-49 when diagnosis (YOCRC group)
* Never received any CRC-related treatment (YOCRC group)
* No CRC confirmed by colonoscopy or pathology (non-YOCRC group)
* Age at 18-49 (non-YOCRC group)

Exclusion Criteria:

* Hospital stay less than 24 hours or with incomplete Complete Blood Count
* Patients with inflammatory bowel disease or hereditary CRC syndromes
* History of other types of primary malignant tumor and other reasons that made them unsuitable for enrollment

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population we extracted in this study were from department of Gastroenterology, department of Oncology, etc. More specifically, there were two major sources for the study participants: some individuals included in our study had relevant symptoms (such as chronic abdominal pain, altered bowel habit, unexplained weight loss, hematochezia), and they received colonoscopy examination under the advice of the doctor, while some individuals come to the hospital just for a comprehensive physical examination (the physical examination items include colonoscopy).
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
The performance of machine learning screening models | through study completion, an average of 1 year
  The performance of young-onset colorectal cancer screening models will be assessed by calculating the area under the receiver operating characteristic (ROC) curve (AUC), Accuracy, Recall, Specificity, Negative predictive value (NPV), Positive predictive value (PPV, or called Precision).

CONTACTS AND LOCATIONS:
Overall Officials: Dong Weiguo, PhD, Study Chair — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
Involving patient privacy information

REFERENCES:
- [Derived] Zhen J, Li J, Liao F, Zhang J, Liu C, Xie H, Tan C, Dong W. Development and validation of machine learning models for young-onset colorectal cancer risk stratification. NPJ Precis Oncol. 2024 Oct 22;8(1):239. doi: 10.1038/s41698-024-00719-2. PMID 39438621